CLINICAL TRIAL: NCT04493580
Title: Effectiveness of Delivering Dialectical Behavioral Therapy Techniques by E-mail in Patients With Borderline Personality Disorder
Brief Title: DBT Techniques by E-mail for Patients With BPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Nazanin Alavi (Other)
Collaborators: Online PsychoTherapy Clinic (Other)
Responsible Party: Sponsor-Investigator, Dr. Nazanin Alavi, Principal Investigator, Assistant Professor, Queen's University
Organization: Queen's University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSIY-391-13
Record Dates: First submitted 2020-07-21; First posted 2020-07-30 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Borderline Personality Disorder
Keywords: Borderline Personality Disorder; Treatment; Barriers to Treatment; Psychotherapy; Dialectal Behavioural Therapy; Online
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Intervention Model Description: Individuals who were referred to the Personality Disorders Service in Kingston, Ontario, Canada, with a diagnosis of BPD by a psychiatrist or family physician were offered the opportunity to either select in-person DBT skills-building program groups (MPE) or an online format of the program (iDBT).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iDBT Treatments (Experimental): 15 weekly DBT sessions. During each session, participants will be sent 30-40 PowerPoint slides including general information on particular topic, overview of skills, and homework sheets to be completed and returned to therapists. Therapists involved will be a psychiatry resident, a psychologist, and a registered nurse who will also facilitate the in-person groups. The content and format of the online program will directly corresponded with that of the in-person group. Participants will be asked to send their homework sheets back to therapists by a specific day each week. The following day, the therapist will email feedback regarding the homework submitted and send next week's PowerPoint slides, information sheets, and homework. In order to be eligible to receive the materials, participants are required to send in homework prior to deadline. If homework was not returned, reminder email will be sent. If more than two sessions are missed, participants are excluded from the program.
  Interventions: Behavioral: iDBT
- In-Person DBT Treatments (Active Comparator): Weekly skills-building groups titled Managing Powerful Emotions (MPE) includes Mindfulness, Distress Tolerance, Emotion Regulation, and Interpersonal Effectiveness. Personality Disorders Service offers more advanced therapy groups for individuals who have successfully completed MPE and wish to continue seeking treatment modalities. Chrysalis Day Treatment Program (CDTP) is for an individual who has progress through two prior phases. In phase one, individuals will participate in a DBT-informed skill-building group (MPE). Once completed, the individual will progress to phase two which includes attending a psychotherapy group, incorporating DBT skills-building. Finally, in phase three, individuals who wish to participate in a more advanced and complex psychological treatment program, apply to participate in CDTP. The CDTP is an intensive day treatment program integrating DBT skills-building, psychodynamic psychotherapy, and a range of other group therapy modalities.
  Interventions: Behavioral: In-Person DBT

INTERVENTIONS:
Behavioral: iDBT — Electronic DBT sessions designed to mirror in-person DBT.
  Arms: iDBT Treatments
Behavioral: In-Person DBT — In-person DBT
  Arms: In-Person DBT Treatments

SUMMARY:
Purpose: The aim of the current study was to evaluate the efficacy of online Dialectical Behavioural Therapy (e-DBT) in the treatment of individuals with symptoms of borderline personality disorder (BPD). Method: Study participants diagnosed with BPD were offered treatment options of either online or in-person format of a DBT skills-building program. During each session, participants were provided with both the material and feedback regarding their previous week's homework. e-DBT protocol and content was designed to mirror in-person content. Participants were assessed by using a Self-Assessment Questionnaire (SAQ) and Difficulties in Emotion Regulation Scale (DERS).

DETAILED DESCRIPTION:
Dialectal Behavioural Therapy: Since 1995, the Personality Disorders Service in Kingston, Ontario, Canada, has developed psychotherapeutic programs that have integrated a range of modalities for the treatment of individuals presenting with borderline personality disorders. Currently, a range of therapy groups is offered, including a weekly skills-building group that is structured to offer the basic DBT curriculum, titled Managing Powerful Emotions (MPE). This MPE curriculum includes Mindfulness, Distress Tolerance, Emotion Regulation, and Interpersonal Effectiveness. MPE has been offered since 2000 as a first-line treatment for individuals who are diagnosed with BPD. The Personality Disorders Service offers more advanced therapy groups for individuals who have completed the MPE and wish to continue seeking treatment modalities. One of the most intensive therapy programs offered is the Chrysalis Day Treatment Program (CDTP). To participate in the CDTP, an individual must progress through two prior phases. In phase one, individuals will participate in a DBT-informed skill-building group (MPE). Once completed, the individual will progress to phase two which includes attending a psychotherapy group, incorporating DBT skills-building. Finally, in phase three, individuals who wish to participate in a more advanced and complex psychological treatment program, apply to participate in CDTP. The CDTP is an intensive day treatment program integrating DBT skills-building, psychodynamic psychotherapy, and a range of other group therapy modalities. This integrated form of psychotherapy is extremely effective, especially for individuals suffering from more severe and prolonged symptomatology and trauma histories.

Recruitment: Individuals who were referred to the Personality Disorders Service in Kingston, Ontario, Canada, with a diagnosis of BPD by a psychiatrist or family physician were offered the opportunity to either select in-person DBT skills-building program groups (MPE) or an online format of the program (iDBT). Inclusion criteria included participants being between the ages of 18 and 65 years at study inception, a diagnosis of borderline personality disorder according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) guidelines. Moreover, participants were required to have the competence to consent and participate, the ability to speak and read English, and have consistent and reliable access to the internet. Participants were excluded from the study if they were experiencing acute hypomanic or manic episodes, acute psychosis, severe alcohol or substance use disorder, or were currently receiving DBT. Individuals who were referred to the program were provided with an information sheet about the study comparing the effectiveness of online treatment to in-person treatment, and those who consented were included in the study. The in-person group served as a control group.

Measurement Scales: Each individual participating in the study completed a pre- and post-program Self-Assessment Questionnaire (SAQ) and Difficulties in Emotion Regulation Scale (DERS) (Weiss, Gratz, & Lavender, 2015). The DERS is a self-report tool designed to obtain an overall measure of the difficulty respondents have with various aspects of emotion regulation. The DERS not only provides an overall score of difficulties with emotion regulation but assesses the following six specific factors related to emotion dysregulation: non-acceptance (non-acceptance of emotional responses), goals (difficulty engaging in goal-oriented behaviours), impulse (difficulty controlling impulses), awareness (lack of emotional awareness), strategies (lack of access to emotion regulation strategies) and clarity (lack of emotional clarity). It was explained to all participants on the consent form and also as part of the first session of both the in-person and electronic groups that the program was created for helping individuals to learn useful skills and strategies for managing their emotions and behaviours, and that it was not a crisis service. iDBT participants were informed that their online therapist would read their emails once a week and thus would not be in a position to respond to crises, such as suicidal impulses or behaviours. Participants were informed that in the case of an emergency, they were to either attend their local emergency department, call emergency services, or call their local crisis line.

Therapy Programs: The therapy program had a duration of 15 weeks, with one DBT session per week. During each online session, participants were individually sent approximately 30-40 PowerPoint slides. These slides included general information on a particular topic, an overview of skills related to the issue being covered, and homework sheets to be completed and returned to their therapists. Therapists involved were a psychiatry resident, a psychologist, and a registered nurse who also facilitated the in-person groups. The content and format of the online program directly corresponded with that of the in-person group. Participants in the online program were asked to send their homework sheets back to the therapists by a specific day each week. The following day, the therapist would email individualized feedback regarding the homework submitted and send the next week's PowerPoint slides, information sheets, and homework. To be eligible to receive the next week's materials, participants were required to send in their homework before the deadline. If the homework was not returned, a reminder email was sent. If more than two sessions were missed, participants were excluded from the program.

Ethical Considerations and Confidentiality: Only the therapists involved in the patients' care had access to the participants' information. The data for variables under study were entered anonymously into a database separate from the clinical file. This study was approved by the Research and Ethics Board of Queen's University, Canada.

ELIGIBILITY:
Inclusion Criteria:

* Borderline Personality Disorder Diagnosis via DSM-5 Guidelines
* Competence to consent and participate
* Ability to speak and read English
* Consistent and reliable access to the internet

Exclusion Criteria:

* Acute hypomanic/manic episodes
* Acute psychosis
* Severe alcohol or substance use disorder
* Currently receiving DBT

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Self-Assessment Questionnaire (SAQ) Changes | Week 1, Week 15
  Self assessment questionnaire
Difficulties in Emotion Regulation Scale (DERS) Changes | Week 1, Week 15
  Self-report tool designed to obtain an overall measure of the difficulty respondents have with various aspects of emotion regulation. The DERS not only provides an overall score of difficulties with emotion regulation, but assesses the following six specific factors related to emotion dysregulation: non-acceptance (non-acceptance of emotional responses), goals (difficulty engaging in goal-oriented behaviors), impulse (difficulty controlling impulses), awareness (lack of emotional awareness), strategies (lack of access to emotion regulation strategies) and clarity (lack of emotional clarity).

CONTACTS AND LOCATIONS:
Overall Officials: Nazanin Alavi, Principal Investigator — Queen's University
Locations (1):
- Hotel Dieu Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Only the therapists involved in the patients' care had access to the participants' information. The data for variables under study were entered anonymously into a database separate from the clinical file. This study was approved by the Research and Ethics Board of Queen's University, Canada.

REFERENCES:
- [Derived] Alavi N, Stephenson C, Rivera M. Effectiveness of Delivering Dialectical Behavioral Therapy Techniques by Email in Patients With Borderline Personality Disorder: Nonrandomized Controlled Trial. JMIR Ment Health. 2021 Apr 30;8(4):e27308. doi: 10.2196/27308. PMID 33835936
- See also: Related Info — https://mental.jmir.org/2021/4/e27308